CLINICAL TRIAL: NCT05590910
Title: The Effects of a Music Intervention on Stress, Anxiety, and Academic Performance Among New Undergraduate Nursing Students
Brief Title: The Effects of a Music Intervention on Stress, Anxiety and Academic Performance on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC20210672H
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2023-11

CONDITIONS: Stress
Keywords: Music, anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: A randomized controlled approach will explore the effects music has on stress and anxiety levels and academic performance among undergraduate nursing students.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention Group (Experimental): The music intervention group will receive a 15-minute music intervention and variables such as heart rate, blood pressure, anxiety, and academic performance will be measured.
  Interventions: Other: Music
- Non-Music Control Group (No Intervention): Variables such as heart rate, blood pressure, anxiety, and academic performance will be measured.

INTERVENTIONS:
Other: Music — Fifteen minutes of classical music will be played overhead in the classroom. The students will be instructed not to use other electronic devices such as ear buds or phones during this time.
  Other Names: Classical music
  Arms: Music Intervention Group

SUMMARY:
This study is examining the effect of listening to music on personal variables such as stress, anxiety, and academic performance. Previous research has shown that listening to music can help in reducing the effects of anxiety and stress.

DETAILED DESCRIPTION:
Students will be divided and randomized into two recording groups: 1.) Music Intervention Group, 2.) Non-Music Control Group. The music intervention group will receive a 15-minute music intervention and variables such as heart rate, blood pressure, anxiety, and academic performance will be measured. The non-music control group will not receive the intervention; however, the same variables will be measured.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Enrolled at UT Health San Antonio School of Nursing clinical course
* First semester undergraduate nursing student

Exclusion Criteria:

* Under 18 years
* Second, third or fourth semester undergraduate nursing student

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Non-Binary
Enrollment: 89 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorgie A Contreras, MSN, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other faculty and published in a peer reviewed journal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared at close of study and after data analysis is completed.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Music Intervention Group | Non-Music Control Group
Started | 49 | 40
Completed | 49 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Music Intervention Group | Non-Music Control Group | Total
Number analyzed (Participants) | 49 | 40 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.55 (6.63) | 24.75 (4.47) | 26.29 (5.73)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Participants Self-Identified as 70 females, 18 males, and 1 non-binary student
  Participants
    Male | 11 | 7 | 18
    Female | 37 | 33 | 70
    Non-Binary | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 19 | 37
  Not Hispanic or Latino | 27 | 18 | 45
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 6 | 12
  White | 35 | 25 | 60
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 18 | 19 | 37
  White | 17 | 6 | 23
  Black or African American | 6 | 6 | 12
  Asian | 4 | 5 | 9
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Other/Mixed | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 40 | 89

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Measurement
Description: Heart rate will be measured using a smartwatch Time 1 (pre-intervention) Time 2 (post-intervention) Time 3 (post-skill)
Time Frame: Baseline (pre-intervention), Time 2 (post intervention, approximately 30 minutes from baseline) and study end (approximately 45 minutes from baseline)
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Music Intervention Group | Non-Music Control Group
Number analyzed (Participants) | 49 | 40
beats per minute
  Time 1 | 83.45 (11.75) | 82.80 (11.92)
  Time 2 | 81.88 (11.82) | 84.38 (10.87)
  Time 3 | 89.31 (13.61) | 91.13 (14.71)

2. Primary Outcome: Blood Pressure Measurement
Description: Change in Blood pressure will be measured using a smartwatch. Only MAP reported: the average arterial pressure throughout one cardiac cycle, systole, and diastole Time 1 Time 2 Time 3
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Music Intervention Group | Non-Music Control Group
Number analyzed (Participants) | 49 | 40
mmHg
  Time 1 | 91.88 (4.82) | 91.39 (5.85)
  Time 2 | 91.14 (4.69) | 90.89 (6.40)
  Time 3 | 93.28 (3.99) | 92.08 (4.21)

3. Primary Outcome: State Trait Anxiety Inventory (STAI)
Description: Change in score on the STAI survey, a 20 item survey with each item rated on a 4 point scale from "almost never" to "almost always. Possible range of scores are from 20-80 with a higher score indicating greater anxiety.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: STAI Scores
Arm/Group | Music Intervention Group | Non-Music Control Group
Number analyzed (Participants) | 49 | 40
STAI Scores
  Time 1 | 43.84 (10.69) | 43.77 (10.04)
  Time 2 | 36.92 (12.81) | 41.63 (12.96)
  Time 3 | 37.51 (11.36) | 38.38 (11.62)

4. Primary Outcome: Academic Performance
Description: Measuring the Skills Competency Recording Performance (Pass/Fail basis)
Time Frame: Baseline to study end (approximately 45 minutes from baseline)
Measure: Number; unit: participants
Arm/Group | Music Intervention Group | Non-Music Control Group
Number analyzed (Participants) | 49 | 40
participants
  Pass | 36 | 26
  Fail | 13 | 14

ADVERSE EVENTS:
Time Frame: approximately 45 minutes
Description: Non-invasive measurements were obtained
Arm/Group | Music Intervention Group | Non-Music Control Group
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/40
Other Adverse Events (participants affected / at risk) | 0/49 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT05590910/Prot_SAP_000.pdf